CLINICAL TRIAL: NCT01580410
Title: A Multi-Center, Open-Label, Randomized Phase II Trial to Evaluate Hematologic Toxicities After HIPEC With Oxaliplatin or Mitomycin C in Patients With Appendiceal Tumors
Brief Title: Surgery and Oxaliplatin or Mitomycin C in Treating Patients With Tumors of the Appendix
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00009326; NCI-2009-00947 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 59109 (Other: Wake Forest University Health Sciences); NCT00904267 (obsolete NCT alias)
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Results first posted 2018-03-21 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Carcinoma of the Appendix; Primary Peritoneal Cavity Cancer
MeSH Terms: conditions — Appendiceal Neoplasms | interventions — Mitomycin; Oxaliplatin; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (mitomycin C) (Experimental): Patients undergo surgical cytoreduction and receive mitomycin C by HIPEC.
  Interventions: Drug: mitomycin C; Procedure: therapeutic conventional surgery; Other: quality-of-life assessment; Drug: hyperthermic intraperitoneal chemotherapy
- Arm II (oxaliplatin) (Experimental): Patients undergo surgical cytoreduction and receive oxaliplatin by HIPEC.
  Interventions: Drug: oxaliplatin; Procedure: therapeutic conventional surgery; Other: quality-of-life assessment; Drug: hyperthermic intraperitoneal chemotherapy

INTERVENTIONS:
Drug: mitomycin C — Given by HIPEC
  Other Names: MITC; MITO; MITO-C; Mitocin-C; MTC
  Arms: Arm I (mitomycin C)
Drug: oxaliplatin — Given by HIPEC
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
  Arms: Arm II (oxaliplatin)
Procedure: therapeutic conventional surgery — Undergo surgery
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Drug: hyperthermic intraperitoneal chemotherapy — Undergo HIPEC

SUMMARY:
This randomized phase II trial is studying the side effects and how well giving oxaliplatin or mitomycin C directly into the abdomen after surgery works in treating patients with tumors of the appendix. Drugs used in chemotherapy, such as oxaliplatin and mitomycin C, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Heating a chemotherapy solution and infusing it directly into the abdomen may kill more tumor cells. Giving these treatments after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the toxicity profiles within 4 weeks of surgery of oxaliplatin and mitomycin C delivered via Hyperthermic Intraperitoneal Chemotherapy in patients with peritoneal surface malignancies from primary appendiceal tumors.

SECONDARY OBJECTIVES:

I. To compare the time to progression in patients treated with oxaliplatin vs. mitomycin C delivered via Hyperthermic Intraperitoneal Chemotherapy for surface malignancies from primary appendiceal tumors.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients undergo surgical cytoreduction and receive mitomycin C by hyperthermic intraperitoneal chemotherapy (HIPEC).

Arm II: Patients undergo surgical cytoreduction and receive oxaliplatin by HIPEC.

After completion of study treatment, patients are followed up at 6, 12, 18, 24, 30, and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed peritoneal surface malignancies from primary appendiceal tumors
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count >= 1,500/mcL
* Platelets >=100,000/mcL
* Total bilirubin =< 1.5 mg/dL
* Creatinine =< 2.0 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 X institutional upper limit of normal
* Alkaline phosphatase =< 3 X institutional upper limit of normal
* Patients must be recovered from both the acute and late effects of any prior surgery, radiotherapy, or other antineoplastic therapy
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or double-barrier method of birth control; abstinence) for the duration of study participation and for 90 days following HIPEC
* Ability to understand and the willingness to sign a written informed consent document (either directly or via a legally authorized representative)
* Participants who have received oxaliplatin during prior systemic chemotherapy regimens are eligible for enrollment in this protocol

Exclusion Criteria:

* Patients with an active infection or with a fever >= 101.3 degrees Fahrenheit (F) within 3 days of the first scheduled day of protocol treatment
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 30 days of HIPEC (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication)
* Patients with carcinoid tumors
* Patients with active central nervous system (CNS) metastases
* Patients with known hypersensitivity to any of the components of oxaliplatin or mitomycin C
* History of prior malignancy within the past 5 years, except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or localized prostate cancer with a current prostate-specific antigen (PSA) of < 1.0 mg/dL on 2 successive evaluations, at least 3 months apart, with the most recent evaluation no more than 4 weeks prior to entry
* Patients who received radiotherapy to more than 25% of their bone marrow
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant/nursing women are excluded from this study because oxaliplatin is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with oxaliplatin, breastfeeding should be discontinued if the mother is treated with oxaliplatin or mitomycin C
* Known human immunodeficiency virus (HIV), hepatitis B or C-positive patients (active, previously treated or both)
* Peripheral neuropathy >= grade 2
* History of allogenic transplant
* History of prior HIPEC
* Evidence of metastatic disease outside of the abdomen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2009-05; Primary Completion 2015-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Levine, Principal Investigator — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Mitomycin C) | Arm II (Oxaliplatin)
Started | 68 | 68
Completed | 57 | 60
Not Completed | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Mitomycin C) | Arm II (Oxaliplatin) | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 48 | 94
  >=65 years | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (12.9) | 55.0 (14.0) | 55.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 40 | 75
  Male | 33 | 28 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 64 | 65 | 129
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 63 | 62 | 125
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 68 | 68 | 136

OUTCOME MEASURES:

1. Primary Outcome: The Difference in the Number of Grade 3 or 4 Hematologic Toxicities (Leukopenia, Thrombocytopenia, and Neutropenia) Between the Mitomycin C and Oxaliplatin Treatments
Description: If a patient has a grade 3 or 4 standard hematologic toxicity (leukopenia, thrombocytopenia, and neutropenia), the patient will be considered to be an event. The observed rates of the 2 treatments will be the primary outcome, and the rates will be analyzed using a 2-sided chi-square test.
Time Frame: Within 4 weeks of surgery
Measure: Number; unit: number of patients with toxicities
Arm/Group | Arm I (Mitomycin C) | Arm II (Oxaliplatin)
Number analyzed (Participants) | 61 | 59
number of patients with toxicities | 8 | 5

2. Secondary Outcome: The Difference in Percentage of Disease-free Survival Between the Two Treatment Arms up to 3 Years
Time Frame: Time to first progression unless the patient's resection status is R2b or 2c, regardless of toxicity or response to study drug, assessed up to 3 years
Measure: Mean (Standard Error); unit: disease-free survival rate (%)
Arm/Group | Arm I (Mitomycin C) | Arm II (Oxaliplatin)
Number analyzed (Participants) | 57 | 53
disease-free survival rate (%) | 61.6 (8.1) | 59.4 (8.1)

3. Secondary Outcome: The Difference in Percentage of Overall Survival Between the Two Treatment Arms up to 3 Years
Time Frame: Interval between surgery and death or date of last contact, assessed up to 3 years
Measure: Mean (Standard Error); unit: overall survival rate (%)
Arm/Group | Arm I (Mitomycin C) | Arm II (Oxaliplatin)
Number analyzed (Participants) | 57 | 53
overall survival rate (%) | 75.7 (6.4) | 79.3 (5.7)

4. Secondary Outcome: Quality of Life as Assessed by Functional Assessment of Cancer Therapy: General (FACT-G)
Description: The FACT-G (Functional Assessment of Cancer Therapy - General) consists of 27 core items assessing patient well-being in four components: Physical (7 items), Social/Family (7 items), Emotional (6 items), and Functional (7 items). Items are rated on a five-point scale: 0-"not at all", 1- "a little bit", 2-"somewhat", 3- "quite a bit" and 4-"very much". The score of each component is the mean times the number of items in the component. The range of the physical, social/family, and functional components I 0-28 and the range of the emotional component is 0-24. The sum of the component scores creates the overall score which has a range of 0-108. For all component scores and overall score, the higher the score the better the QOL.
Time Frame: Throughout study completion, up to 3 years
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I (Mitomycin C) | Arm II (Oxaliplatin)
Number analyzed (Participants) | 57 | 53
units on a scale | 85.5 (1.6) | 89.6 (1.7)

ADVERSE EVENTS:
Arm/Group | Arm I (Mitomycin C) | Arm II (Oxaliplatin)
All-Cause Mortality (participants affected / at risk) | 1/58 | 1/61
Serious Adverse Events (participants affected / at risk) | 51/58 | 54/61
Other Adverse Events (participants affected / at risk) | 58/58 | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Mitomycin C) (N=58) | Arm II (Oxaliplatin) (N=61)
Low WBC (Investigations) | 3 (3) | 2 (2)
low Platelets (Investigations) | 1 (1) | 3 (4)
Low Hemoglobin (Investigations) | 35 (35) | 36 (36)
Nausea (Gastrointestinal disorders) | 7 (7) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 9 (9)
Anorexia (General disorders) | 10 (10) | 8 (8)
Obstruction, GI: Small bowel (Gastrointestinal disorders) | 1 (1) | 1 (1)
Creatinine (Investigations) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 14 (14)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (8)
Hypotension (Cardiac disorders) | 2 (2) | 3 (3)
Low ANC (Investigations) | 1 (1) | 4 (4)
Fatigue (General disorders) | 6 (6) | 7 (7)
Weight loss (General disorders) | 4 (4) | 2 (2)
hyperglycemia (Investigations) | 3 (3) | 6 (6)
hypocalcemia (Investigations) | 1 (1) | 0 (0)
hyponatremia (Investigations) | 3 (3) | 2 (2)
hypokalemia (Investigations) | 7 (7) | 1 (1)
hypoalbuminemia (Investigations) | 16 (16) | 19 (19)
hyperbilirubinemia (Investigations) | 1 (1) | 0 (0)
serum glutamic pyruvic transaminase (Investigations) | 12 (12) | 9 (9)
hypophosphatemia (Investigations) | 13 (13) | 14 (14)
serum glutamic oxaloacetic transaminase (Investigations) | 16 (16) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 5 (5)
Confusion (General disorders) | 1 (1) | 1 (1)
Mood alteration: Agitation (General disorders) | 4 (4) | 2 (2)
Anxiety (General disorders) | 1 (1) | 2 (2)
Depression (General disorders) | 1 (1) | 1 (1)
Pain: Abdomen (General disorders) | 5 (5) | 4 (4)
Acidosis (Investigations) | 2 (2) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2)
Infection Bladder (Infections and infestations) | 1 (1) | 1 (1)
creatine phosphokinase (Investigations) | 1 (1) | 0 (0)
Pain: Chest/thorax (General disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
disseminated intravascular coagulation (Investigations) | 1 (1) | 0 (0)
Prolonged QTc interval (Investigations) | 1 (1) | 0 (0)
functional obstruction of bowel (Gastrointestinal disorders) | 8 (8) | 10 (10)
Lymphopenia (Investigations) | 20 (21) | 25 (28)
Malabsorption (Gastrointestinal disorders) | 2 (2) | 4 (4)
Death not associated with CTCAE term: Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Pain: Muscle (General disorders) | 2 (2) | 3 (3)
infection associated with Lymphopenia (Infections and infestations) | 1 (1) | 1 (1)
Pain: Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 9 (9) | 10 (11)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
International Normalized Ratio of prothrombin time (Investigations) | 1 (1) | 0 (0)
Pain: Scrotum (General disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Urinary with low grade neutropenia (Infections and infestations) | 2 (2) | 0 (0)
Mental status (General disorders) | 1 (1) | 0 (0)
Hemorrhage, GI: Lower GI (Vascular disorders) | 2 (2) | 1 (1)
Hemorrhage/bleeding associated with surgery, intra-operative or postoperative (Vascular disorders) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: Abdomen (Infections and infestations) | 3 (3) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils: Peritoneal cavity (Infections and infestations) | 2 (2) | 2 (2)
Cardiac troponin I (Investigations) | 1 (1) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fistula, GI: Abdomen (Gastrointestinal disorders) | 2 (2) | 0 (0)
Leak (including anastomotic), GI: Leak (Gastrointestinal disorders) | 1 (1) | 1 (1)
Leak (including anastomotic), GI: Small bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Necrosis, GI: Small bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lung Infection with high grade neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: Pelvis (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: Wound (Infections and infestations) | 1 (1) | 1 (1)
Infection with unknown ANC: Peritoneal cavity (Infections and infestations) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy): Left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Prolonged intubation after pulmonary resection (>24 hrs after surgery) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Infection with high grade neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Blood Infection with high grade neutropenia (Infections and infestations) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Mitomycin C) (N=58) | Arm II (Oxaliplatin) (N=61)
Low WBC (Investigations) | 11 (11) | 22 (22)
low Platelets (Investigations) | 33 (33) | 27 (27)
Low Hemoglobin (Investigations) | 22 (22) | 22 (22)
Nausea (Gastrointestinal disorders) | 19 (19) | 18 (18)
Vomiting (Gastrointestinal disorders) | 24 (24) | 17 (17)
Diarrhea (Gastrointestinal disorders) | 18 (18) | 8 (8)
Anorexia (General disorders) | 20 (20) | 19 (19)
Alkaline phosphatase (Investigations) | 31 (31) | 27 (27)
Creatinine (Investigations) | 2 (2) | 2 (2)
Proteinuria (Investigations) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 10 (10)
Hypertension (General disorders) | 2 (2) | 3 (3)
Hypotension (Cardiac disorders) | 8 (8) | 4 (4)
Neuropathy: sensory (Cardiac disorders) | 6 (7) | 1 (1)
Low ANC (Investigations) | 2 (2) | 3 (3)
Taste alteration (General disorders) | 4 (4) | 4 (4)
Insomnia (General disorders) | 11 (11) | 5 (5)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rigors/chills (General disorders) | 1 (1) | 1 (1)
Sweating (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 30 (30) | 22 (22)
Weight loss (General disorders) | 26 (26) | 34 (34)
hyperglycemia (Investigations) | 42 (42) | 42 (42)
hypocalcemia (Investigations) | 3 (3) | 4 (4)
hypomagnesemia (Investigations) | 8 (8) | 6 (6)
hyponatremia (Investigations) | 35 (35) | 29 (29)
hypokalemia (Investigations) | 26 (26) | 31 (31)
Bicarbonate serum-low (Investigations) | 2 (2) | 0 (0)
hypoalbuminemia (Investigations) | 33 (33) | 35 (35)
hyperbilirubinemia (Investigations) | 2 (2) | 4 (4)
serum glutamic pyruvic transaminase (Investigations) | 31 (31) | 37 (37)
hypophosphatemia (Investigations) | 5 (5) | 6 (6)
Constipation (Gastrointestinal disorders) | 6 (6) | 4 (4)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2) | 1 (1)
serum glutamic oxaloacetic transaminase (Investigations) | 31 (31) | 43 (43)
hypermagnesemia (Investigations) | 2 (2) | 1 (1)
hyperkalemia (Investigations) | 2 (2) | 4 (4)
hypernatremia (Investigations) | 2 (2) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Dysphagia (General disorders) | 1 (1) | 0 (0)
Fever without neutropenia (General disorders) | 6 (6) | 5 (5)
Constitutional Symptoms - Other (General disorders) | 1 (1) | 0 (0)
Cardiac Arrhythmia - Other (Cardiac disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Edema: limb (Vascular disorders) | 2 (2) | 3 (3)
Edema: trunk/genital (General disorders) | 1 (1) | 1 (1)
Edema: viscera (Vascular disorders) | 3 (3) | 1 (1)
Dehydration (General disorders) | 2 (2) | 2 (2)
Confusion (General disorders) | 2 (2) | 0 (0)
Mood alteration: Agitation (General disorders) | 1 (1) | 0 (0)
Anxiety (General disorders) | 5 (5) | 4 (4)
Depression (General disorders) | 1 (1) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Distension bloating, abdominal (General disorders) | 4 (4) | 1 (1)
Pain: Abdomen (General disorders) | 8 (8) | 18 (18)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pain: Joint (General disorders) | 2 (2) | 1 (1)
Ascites (non-malignant) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 16 (16)
Conduction abnormality/atrioventricular heart block (Cardiac disorders) | 1 (1) | 0 (0)
Pain: Back (General disorders) | 2 (2) | 0 (0)
Infection Bladder (Infections and infestations) | 1 (1) | 1 (1)
Pain Bladder (General disorders) | 1 (1) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Wound complication, non-infectious (General disorders) | 10 (10) | 8 (8)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hiccoughs (hiccups, singultus) (General disorders) | 2 (2) | 1 (1)
hypertriglyceridemia (Investigations) | 1 (1) | 0 (0)
functional obstruction of bowel (Gastrointestinal disorders) | 5 (5) | 4 (4)
Watery eye (epiphora, tearing) (Eye disorders) | 1 (1) | 0 (0)
Lymphopenia (Investigations) | 24 (24) | 21 (21)
Pain: Muscle (General disorders) | 4 (4) | 5 (5)
Pain: Neuralgia/peripheral nerve (General disorders) | 1 (1) | 0 (0)
Pain Oral cavity (General disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
International Normalized Ratio of prothrombin time (Investigations) | 1 (1) | 1 (1)
Supraventricular and nodal arrhythmia: Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 9 (9) | 5 (5)
Pain: Stomach (General disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia: Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 3 (3)
Pain: Urethra (General disorders) | 1 (1) | 0 (0)
Urinary with low grade neutropenia (Infections and infestations) | 1 (1) | 1 (1)
Hemorrhage GU: Urinary (Vascular disorders) | 3 (3) | 2 (2)
Leak (including anastomotic), GI: Pancreas (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1) | 0 (0)
Cognitive disturbance (General disorders) | 1 (1) | 1 (1)
Leak (including anastomotic), GI: Leak (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis/stomatitis Oral cavity (Infections and infestations) | 1 (1) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils: Wound (Infections and infestations) | 2 (2) | 1 (1)
Infection with unknown ANC Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Prolonged chest tube drainage or air leak after pulmonary resection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intra-operative injury: NERVES: Peripheral sensory (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The worst adverse event of each type was recorded for the course of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes